CLINICAL TRIAL: NCT06831292
Title: Molecular Mechanisms for Male Fertility: Can Diet Change Sperm SncRNA and the Reproductive Potential?
Brief Title: The Effects of Diet on Small Non-coding RNA I Sperm Cells and the Possible Effects on Reproductive Success: Diet Intervention Effects on Sperm
Acronym: DIET-IS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Susanne Liffner, Principal Investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RÖ-961659 substudy 3
Record Dates: First submitted 2024-09-17; First posted 2025-02-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Changes in SncRNA in Sperm; Male Fertility; RNA Profile
Keywords: male fertility; small non-coding RNA; diet; infertility; reproduction; diet intervention
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet intervention- Nordic nutrition recommendations (Active Comparator): The intervention group will receive groceries with planned recipes during the hormonal treatment period for the woman (11-14 days) before IVF. The meal plan will be according to the Nordic dietary guidelines and individualized to match total energy expenditure.
  Interventions: Dietary Supplement: Diet intervention NMR
- No diet intervention (No Intervention): No intervention - this group will only receive standard care

INTERVENTIONS:
Dietary Supplement: Diet intervention NMR — Participants will receive groceries to their homes with planned recipes. The recipes are planned by using the Nordic nutrition councils recommendations.
  Arms: Diet intervention- Nordic nutrition recommendations

SUMMARY:
In this study, patients with infertility treated with IVF at the Center of Reproductive Medicine in Linköping, Sweden, will receive recipes and food according to Nordic dietary guidelines. The purpose is to investigate whether a short diet intervention is sufficient to improve sperm quality and shift the small non-coding RNA profile. In our previous study sperm showed rapid response to diet.

DETAILED DESCRIPTION:
This study is a randomized controlled trial recruiting males seeking IVF treatment with their female partner at the Center for Reproductive Medicine in Linkoping, Sweden. Men will be randomized to a control group or diet intervention group.

The intervention group will receive groceries with planned recipes during the hormonal treatment period for the woman (11-14 days) before IVF. The meal plan will be according to the Nordic dietary guidelines and individualized to match total energy expenditure.

The male partner must accept to participate in the diet intervention in order to be included and the female partner can choose to participate in the diet intervention but it is optional. Sperm samples will be collected before the start of hormonal treatment and on ovum pick-up day. Weight will be measured before and after the intervention. Sperm samples will be processed as standard practice at the fertility clinic. Sperm samples will be used for molecular analysis, such as small RNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Male (biological) partner in infertile couple, scheduled for first IVF treatment
* Mature sperm cells in semen
* Able to speak and read Swedish
* Omnivore
* Will refrain from nicotine and alcohol during intervention
* Sperm sampled provided no more than 3 weeks before intervention start

Exclusion Criteria:

* Former or present malignant disease
* Former radiotherapy in pelvic area
* Former chemotherapy
* Known genetic/chromosomal disorder
* Food allergy

Ages: 23 Years to 56 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sperm RNA profile changes | At day at ovum pick-up
  Small RNA profiling and sequencing will be performed on sperm cells provided by participant at the start of controlled ovarian hormone stimulation of partner and at time of ovum pick-up and compared between the intervention groups.
Sperm total count | At day of ovum pick-up
  Sperm total count in millions, assessed by sperm analysis
Sperm concentration | At day of ovum pick-up
  Sperm concentration assessed by sperm analysis in millions/ml, with total sperm count in millions, divided by semen volume assessed in ml.
Sperm sample analysis | At day of ovum pick-up
  Sperm motility assessed, proportion of motile sperm to total amount of sperm, reported in percent

SECONDARY OUTCOMES:
Fertilization rate | Day one after ovum pick-up
  Number of normally fertilised oocytes, assessed as proportion of total number of oocytes retrieved (percent)
High quality embryo rate | Day 6 after ovum pick-up
  Number of high quality embryo in relation to total number of oocytes fertilised
Embryos frozen | Day 5 and/or 6 after ovum pick-up
  Number of good quality embryos frozen
Clinical pregnancy rate | Assessed 5-7 weeks after ovum pick-up
  Defined by viable intra-uterine pregnancy at ultrasonography in gestational week 7-9
Pregnancy rate | Assessed three weeks after ovum pick-up
  Positive pregnancy test in urine (hCG) after IVF

OTHER OUTCOMES:
Oxidative stress in sperm sample | At day of ovum pick-up
  Reactive oxygen species analysis of semen

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No